CLINICAL TRIAL: NCT06777979
Title: CD19-CD22-Bispecific Chimeric Antigen Receptor (CAR) T Cell Therapy for Pediatric Patients With Acute Lymphoblastic Leukemia (1922CAR)
Brief Title: CD19-CD22-Bispecific Chimeric Antigen Receptor (CAR) T Cell Therapy for Pediatric Patients With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1922CAR; NCI-2024-10103 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Recurrent Acute Lymphoblastic Leukemia; Recurrent B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — fludarabine; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD19-CD22-CAR T cell therapy (Experimental): This study has two parts:
  Collection and Manufacturing Phase - Patients will have white blood cells collected in the St. Jude Blood Donor Center through a procedure called apheresis, or your doctors may use a previously collected frozen product. The collected cells will be engineered to improve their ability to recognize and kill cancer cells. The final cell product is referred to as the CD19-CD22 CAR T cells.
  Treatment Phase - Eligible patients will receive chemotherapy before receiving the CAR T cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Device: CD19-CD22 CAR T cell infusion

INTERVENTIONS:
Drug: Fludarabine — IV
Drug: Cyclophosphamide — IV
Drug: Mesna — IV
Device: CD19-CD22 CAR T cell infusion — CAR T cell infusion will be given intravenously, either centrally or peripherally.

SUMMARY:
This study is a phase I study designed to evaluate the safety of CD19-CD22-CAR T cells.

Primary Objective:

To determine the safety profile and propose the recommended phase 2 dose (RP2D) of autologous CD19-CD22-CAR T cells in patients ≤ 21 years of age with recurrent/refractory CD19- and/or CD22-positive leukemia.

Secondary Objective:

To evaluate the anti-leukemic activity of CD19-CD22-CAR T cells.

DETAILED DESCRIPTION:
Treatment will include a single course of lymphodepleting chemotherapy (fludarabine/cyclophosphamide) followed by CAR T cell infusion. CAR T cell dose will be determined by the protocol-defined dose escalation scheme, based on the number of CAR+ T cells and participant weight.

ELIGIBILITY:
Collection and Manufacturing Eligibility

Inclusion Criteria:

* Age <21 years old
* Relapsed/refractory CD19- and/or CD22-positive acute leukemia defined as:

  *CD19 and/or CD22-positivity confirmed within 2 months and after receipt of any CD19 or CD22-directed therapy
  * Second or greater relapse
  * Any relapse after allogeneic HCT
  * Refractory disease (primary or in relapse) despite therapy designed to induce remission
* Estimated life expectancy of > 12 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥50 (Appendix A)
* For females of childbearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum or urine pregnancy test within 7 days prior to enrollment

Exclusion Criteria:

* Known primary immunodeficiency
* Known HIV positivity
* Known contraindication to receiving protocol defined lymphodepleting
* chemotherapy regimen
* History of hypersensitivity reaction to murine protein-containing products

Treatment Eligibility

Inclusion Criteria:

* Age < 21 years old
* Detectable disease in the bone marrow
* Estimated life expectancy of > 8 weeks
* Karnofsky or Lansky (age-dependent) performance score > 50 (Appendix A)
* Adequate cardiac function defined as left ventricular ejection fraction >40%, or shortening fraction > 25%
* EKG without evidence of clinically significant arrhythmia
* Adequate renal function defined as creatinine clearance or radioisotope GFR >50 mL/min/1.73m2 (GFR >40 mL/min/1.73m2 if <2 years of age)
* Adequate pulmonary function defined as forced vital capacity (FVC) >50% of predicted value; or pulse oximetry >92% on room air
* Total bilirubin < 3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5 times the upper limit of normal for age
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* Prior to planned CAR T cell infusion, patients with a history of prior allogeneicHCT must be at least 3 months from HCT, have no evidence of acute GVHD, and have not received a donor lymphocyte infusion (DLI) within the 28 daysprior to planned infusion
* For females of childbearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum or urine pregnancy test within 7 days prior to enrollment
  * If sexually active, agreement to use birth control until 3 months after T cell infusion. Male partners should use a condom.

Exclusion Criteria:

* Known primary immunodeficiency
* Known HIV positivity
* Known contraindication to receiving protocol defined lymphodepleting
* chemotherapy regimen
* History of hypersensitivity reactions to murine protein-containing products
* Severe, uncontrolled bacterial, viral or fungal infection
* Active CNS-3 disease
* Evidence of active, uncontrolled neurologic disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of CD19-CD22-CAR T cells | up to 4 weeks after CD19-CD22-CAR T-cell infusion
  Phase I design to determine the RP2D of CD19-CD22-CAR T cells. Two (2) dose levels will be evaluated (1x106 and 3x106cells/kg).
Incidence of adverse events | up to 4 weeks after CD19-CD22-CAR T-cell infusion
  Will be assessed and graded using the CTCAE v5.0, with the exception of CRS and ICANS, which will be graded according to ASTCT Consensus Guidelines. Adverse events will be summarized descriptively and dose limiting toxicity (DLT) rate will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Epperly, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols